CLINICAL TRIAL: NCT06047067
Title: BIOAEROSOL SAMPLING DEVICE (BSD) CLINICAL STUDY: Performance of Respiratory Pathogen Bioaerosol Sampling Device Compared to Matched Swab Sample With Molecular and Antigen Assays That Can Detect SARS-CoV-2 Phase II Validation
Brief Title: Bioaerosol Sampling Device (BSD) Clinical Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cantor BioConnect, Inc. (Network)
Collaborators: 3M (Industry); Biomedical Advanced Research and Development Authority (U.S. Federal Agency); JPRA Enterprises, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: CBC-1051
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: COVID-19; Rapid diagnostic test; SARS-CoV-2; SARS-CoV-1
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Samples to be retained without DNA for 1 year and discarded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical trial is to learn about the bioaerosol sampling device (BSD) and how it can sample patient bioaerosols (breath) and patient's nares for the detection of COVID-19 viral particles in patients seeking to be tested for COVID-19.

DETAILED DESCRIPTION:
SARS-CoV-2, the virus which causes COVID-19, is transmissible through bioaerosols. Routine accessible, non-invasive, sensitive testing could play a role in reducing the spread of the disease and controlling the current and future pandemics. The Bioaerosol Sampling Device may offer both comfort and the potential to increase the ability to detect patients earlier in the infection cycle than a swab. The primary objective of the research is to generate BSD performance data with detection by RT-PCR and at-home molecular and antigen assays, compared to nasal swab comparator detected by EUA or 510k cleared RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

Any patient 5 years or older who wants to be tested Patients may be symptomatic or asymptomatic based on CDC guidelines Patients may be suspected of having COVID-19 based on CDC guidelines Patient's COVID-19 status should be unknown Patients younger than 12 should be assisted by an adult

Exclusion Criteria:

Unable to self-consent Concurrent enrollment in other trials involving same-day nasal cavity sampling

Contraindication to nasal sampling as performed according to the clinical site policies and procedures, including:

Unable to tolerate Nasal Swab Sampling History of perforation of the nasal septum or prone to nosebleed Head or facial injury/surgery within the past 6 months On anticoagulant therapy including anti-platelet therapy Nasal or nasal aspirate and nasal wash performed as standard of care.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient arriving at a participating site wanting to be tested with COVID-19, status unknown. Demographic information will be collected. Best efforts will be made to enroll subjects with diverse socioeconomic and educational obtainment.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-05-19 (Estimated); Study Completion 2024-05-19 (Estimated)

PRIMARY OUTCOMES:
BSD detection of SARS-CoV-2: The primary objective of the research is to generate BSD performance data with detection by RT-PCR and at-home molecular and antigen assays, compared to nasal swab comparator detected by EUA or 510k cleared RT-PCR. | 1 year
  Aim 1 Objective 1: The primary objective of Aim 1 (A1O1) is to generate and evaluate BSD performance data for patients enrolled within the first 3 days of symptoms, with detection by RT-PCR and at-home molecular and antigen assays, compared to Nasal Swab Comparator detected by EUA or 510k cleared RT-PCR assays.
  Aim 1 Objective 2a: The secondary objective (A1O2a) of Aim 1 is to generate and evaluate the same BSD performance data as Aim 1 objective 1, but to do so for patients enrolled within the first 7 days of symptom onset.
  Aim 1 Objective 2b: The secondary objective (A1O2b) of Aim 1 is to generate and evaluate the same BSD performance data as Aim 1 objective 1, but to do so for any patients seeking to get tested for SARS-CoV-2 test, regardless of presence of symptoms or symptom onset.

SECONDARY OUTCOMES:
BSD performance data: Generate and evaluate the performance data evaluated based on virus load. | 1 year
  Aim 2 Objective 1: The primary objective of Aim 2 (A2O1) is to generate and evaluate BSD performance data for enrolled patients, with detection by at-home antigen assays, compared to Nasal Swab Comparator detected by EUA or 510k cleared RT-PCR assays with Ct values of less than 30. This objective will focus will be to evaluate the sensitivity of the BSD to detect SARS-CoV-2 virus with at-home antigen tests among specimens with a nasal swab RT-PCR Ct value of less than 30.
  Aim 2 Objective 2: The secondary objective of Aim 2 (A2O2) is to generate and evaluate BSD performance data for enrolled patients, with detection by PCR, compared to Nasal Swab Comparator detected by EUA or 510k cleared RT-PCR assays, in order to derive a correlation between virus load collected via BSD and virus load collected via nasal swab, both as measured by RT-PCR Ct value on the same RT-PCR assay.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Azurin, MD, Principal Investigator — JPRA Enterprises, LLC
Locations (5):
- United States (5):
  - JPRA Enterprise, LLC, South Gate, California
  - Alfa Medical Research, Hollywood, Florida
  - Alfa Medical Urgent Care, Pembroke Pines, Florida
  - HDH Research, Houston, Texas
  - HDH Research, Humble, Texas

IPD SHARING:
Plan to Share IPD: Undecided
3M governs the policies, procedures and permissions. Submission of data to the FDA is probable.

REFERENCES:
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Background] Wang CJ, Ng CY, Brook RH. Response to COVID-19 in Taiwan: Big Data Analytics, New Technology, and Proactive Testing. JAMA. 2020 Apr 14;323(14):1341-1342. doi: 10.1001/jama.2020.3151. No abstract available. PMID 32125371
- [Background] Mercer TR, Salit M. Testing at scale during the COVID-19 pandemic. Nat Rev Genet. 2021 Jul;22(7):415-426. doi: 10.1038/s41576-021-00360-w. Epub 2021 May 4. PMID 33948037
- [Background] Marra P, Colacurcio V, Bisogno A, De Luca P, Calvanese M, Petrosino M, De Bonis E, Troisi D, Cassandro C, Cavaliere M, Ralli M, Cassandro E, Scarpa A. Evaluation of Discomfort in Nasopharyngeal Swab Specimen Collection for SARS-CoV-2 Diagnosis. Clin Ter. 2021 Sep 29;172(5):448-452. doi: 10.7417/CT.2021.2357. PMID 34625778
- [Background] Obuchowski NA, Zhou XH. Prospective studies of diagnostic test accuracy when disease prevalence is low. Biostatistics. 2002 Dec;3(4):477-92. doi: 10.1093/biostatistics/3.4.477. PMID 12933593
- [Background] Li J, Fine J. On sample size for sensitivity and specificity in prospective diagnostic accuracy studies. Stat Med. 2004 Aug 30;23(16):2537-50. doi: 10.1002/sim.1836. PMID 15287083
- [Background] Jarvis KF, Kelley JB. Temporal dynamics of viral load and false negative rate influence the levels of testing necessary to combat COVID-19 spread. Sci Rep. 2021 Apr 28;11(1):9221. doi: 10.1038/s41598-021-88498-9. PMID 33911131
- [Background] Parmar H, Montovano M, Banada P, Pentakota SR, Shiau S, Ma Z, Saibire K, Chopoorian A, O'Shaughnessy M, Hirsch M, Jain P, Demirdjian G, Karagueuzian M, Robin T, Salvati M, Patel B, Alland D, Xie YL. RT-PCR negative COVID-19. BMC Infect Dis. 2022 Feb 13;22(1):149. doi: 10.1186/s12879-022-07095-x. PMID 35152885
- [Background] Pecoraro V, Negro A, Pirotti T, Trenti T. Estimate false-negative RT-PCR rates for SARS-CoV-2. A systematic review and meta-analysis. Eur J Clin Invest. 2022 Feb;52(2):e13706. doi: 10.1111/eci.13706. Epub 2021 Dec 5. PMID 34741305
- [Background] Kanji JN, Zelyas N, MacDonald C, Pabbaraju K, Khan MN, Prasad A, Hu J, Diggle M, Berenger BM, Tipples G. False negative rate of COVID-19 PCR testing: a discordant testing analysis. Virol J. 2021 Jan 9;18(1):13. doi: 10.1186/s12985-021-01489-0. PMID 33422083
- [Background] Phuphuakrat A, Pasomsub E, Srichatrapimuk S, Kirdlarp S, Suksatu A, Srisaowakarn C, Manopwisedjaroen S, Ludowyke N, Purwono PB, Priengprom T, Wongsa A, Thakkinstian A, Hongeng S, Malathum K, Thitithanyanont A, Tassaneetrithep B. Detectable Duration of Viable SARS-CoV-2, Total and Subgenomic SARS-CoV-2 RNA in Noncritically Ill COVID-19 Patients: a Prospective Cohort Study. Microbiol Spectr. 2022 Jun 29;10(3):e0050322. doi: 10.1128/spectrum.00503-22. Epub 2022 May 23. PMID 35604133